CLINICAL TRIAL: NCT02254057
Title: Tolerability and Pharmacokinetics/-Dynamics of Single Rising Doses of 0.1 mg, 0.3 mg, 1.0 mg, 2.5 mg, 5.0 mg, and 10.0 mg BIBT 986 BS (IV Infusion Over 30 Minutes) in Healthy Male Subjects. Placebo Controlled, Double Blind Randomised at Each Dose Level
Brief Title: Tolerability and Pharmacokinetics/-Dynamics of Single Rising Doses BIBT 986 BS in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1192.1
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy

ARMS (2):
- BIBT 986 BS - single rising dose (Experimental)
  Interventions: Drug: BIBT 986 BS - single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBT 986 BS - single rising dose
  Arms: BIBT 986 BS - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the tolerability of BIBT 986 BS after intravenous infusions of 0.1, 0.3, 1.0, 2.5, 5.0, and 10 mg, to assess the pharmacokinetics of BIBT 986 BS after intravenous infusion and to assess the effect of BIBT 986 BS on blood coagulation parameters

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 55 years
* BMI >= 18.5 and <= 29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Any bleeding disorder including prolonged or habitual bleeding
* History of other hematologic disease, cerebral bleeding (e.g. after a car accident), commotio cerebri
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Seasonal rhinitis
* Thrombocytes < 150000/μl
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 2 months prior to administration or during trial)
* Smoker (> 10 cigarettes or >3 cigars or >3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Use of methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.), grapefruit or grapefruit juice, alcohol, green tea, or tobacco < 5 days prior to administration of study drug or during trial
* Blood donation or loss > 400 ml, < 1 month prior to administration or during the trial
* Excessive physical activities < 5 days prior to administration of study drug or during trial
* Clinically relevant laboratory abnormalities
* Any ECG value outside of the reference range of clinical relevance including, but not limited to QRS interval > 110 ms or QTcB > 450 ms
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2002-07; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single dose administration) | up to 48 hours after start of infusion
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration after single dose administration) | up to 48 hours after start of infusion
C29 (plasma concentration of BIBT 986 BS at the end of infusion) | 29 minutes after start of infusion
t1/2 (Terminal half-life of the analyte in plasma after single dose administration) | up to 48 hours after start of infusion
CL (Total clearance of the analyte in plasma following intravascular administration) | up to 48 hours after start of infusion
Vss (Apparent volume of distribution at steady state following intravascular administration) | up to 48 hours after start of infusion
urinary excretion of BIBT 986 BS | up to 48 hours after start of infusion
CLR (Renal clearance of the analyte in plasma following intravascular administration) | up to 48 hours after start of infusion
MRT (Mean residence time of drug molecules in the body after intravascular administration) | up to 48 hours after start of infusion
Change in activated partial thromboplastin time (aPTT) | up to 48 hours after start of infusion
Change in International Normalised Ratio (INR) | up to 48 hours after start of infusion
Change in ecarin clotting time (ECT) | up to 48 hours after start of infusion
Change in thrombin time (TT) | up to 48 hours after start of infusion
Number of patients with clinically significant findings in vital signs | up to 48 hours after start of infusion
  pulse rate, blood pressure
Number of patients with clinically significant findings in electrocardiogram | up to 48 hours after start of infusion
Number of patients with clinically significant findings in laboratory tests | up to 48 hours after start of infusion
Number of patients with adverse events | up to 48 hours after start of infusion
Number of patients with histamine in blood | up to 48 hours after start of infusion